CLINICAL TRIAL: NCT03856528
Title: Infections of the Central Nervous System - an Observational Cohort Study
Brief Title: Infections of the Central Nervous System
Status: Withdrawn | Type: Observational
Why Stopped: due to personal changes
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01244; me19Sutter2
Record Dates: First submitted 2019-02-26; First posted 2019-02-27 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Adult Patients With Suspected Meningitis and/or Encephalitis
Keywords: meningitis; encephalitis
MeSH Terms: conditions — Meningitis; Encephalitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: collection of patient data — Patient data will be obtained using digital patients records systems. The following data will be assessed: Demographics and baseline patient characteristics (e.g., gender, age, hospital admission and discharge dates), diagnoses, comorbidities (history of meningitis and/or encephalitis, epileptic disorders, remote stroke, remote intracranial bleeding, remote autoimmune disease, neurodegenerative disorders), laboratory features (blood cultures, lumbar puncture), features of neuroimaging (e.g., time admission-to-CT), therapeutic features (incl. time admission-to-treatment), Patients' outcome measures (Glasgow Outcome Score)

SUMMARY:
This study is to describe the incidence of infectious meningitis and/or encephalitis, and to analyze clinical, diagnostic and treatment characteristics of patients with suspected (and subsequently verified and not verified) infection.

DETAILED DESCRIPTION:
The specific aims of the study include:

1. To assess the incidence, the diagnostic workup, and the treatment characteristics of patients with suspected and confirmed ME.
2. To examine clinical differences between patients with initially suspected and confirmed infectious Meningitis (ME) versus those with suspected but not confirmed infectious ME.
3. To evaluate potentially prognostic factors for pathological CT findings (especially expanding cerebral mass lesions) in patients with suspected infectious ME.
4. To identify a specific group of patients that benefit from cranial CT prior to LP.
5. To examine possible complications (e.g., hematoma, postpuncture headache, cerebral herniation, …) of lumbal punction (LP) and their correlations to pathologic signs on cranial CT.
6. To compare the outcome between patients with suspected infectious ME and cranial CT prior to LP versus patients without prior cranial CT.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged ≥18 years admitted to the University Hospital Basel with confirmed infectious meningitis and/or encephalitis as principal and/or secondary diagnosis from January 2006 to December 2021 with or without cranial CT prior to LP
* All patients aged ≥18 years admitted to the University Hospital Basel over the same time period with suspected infectious meningitis and/or encephalitis as principal and/or secondary diagnosis with or without cranial CT

Exclusion Criteria:

* Patients without suspected infectious meningitis and/or encephalitis.
* Patients with the diagnosis of meningitis/encephalitis confirmed prior to hospital admission
* Patients who have refused "General Consent" (i.e., written agreement of patients which allows the further use of their collected medical data for research purposes in encoded form).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the University Hospital Basel with suspected or confirmed infectious meningitis/encephalitis over a 10-year period (from January 2006 to December 2021).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of patients with suspected and confirmed ME (number) | single time point assessment during hospital stay (up to 4 weeks)
  assessment of number of patients with suspected and confirmed ME
Pathologic CT findings | single time point assessment during hospital stay (up to 4 weeks)
  assessment of number of patients with pathologic CT findings
Pathologic CT findings constituting a risk factor for herniation after performance of LP | single time point assessment during hospital stay (up to 4 weeks)
  assessment of number of patients with pathologic CT findings constituting a risk factor for herniation after performance of LP

SECONDARY OUTCOMES:
hematoma (number) | single time point assessment during hospital stay (up to 4 weeks)
  hematoma as a complication of LP
Glasgow Outcome Score | single time point assessment during hospital stay (up to 4 weeks)
  scale of patients with brain injuries that groups victims by the objective degree of recovery.The scale consists of five ordinal outcome categories: good recovery (able to live independently, able to return to work or school), moderate disability (able to live independently, unable to return to work or school), severe disability (able to follow commands, unable to live independently), persistent vegetative state (unable to interact with the environment, unresponsive), and death.
postpuncture headache (number) | single time point assessment during hospital stay (up to 4 weeks)
  postpuncture headache as a complication of LP
cerebral herniation (number) | single time point assessment during hospital stay (up to 4 weeks)
  cerebral herniation as a complication of LP
pathological CT findings (number) | single time point assessment at hospitalisation (Day1)
  number and evaluation of pathological CT findings (especially expanding cerebral mass lesions) in patients with suspected infectious ME
kind of medication | single time point assessment during hospital stay (up to 4 weeks)
  assessment of medication (treatment characteristics ) of patients with suspected and confirmed ME
Intensive Care Delirium Screening Checklist (ICDSC) | single time point assessment during hospital stay (up to 4 weeks)
  The ICDSC is a screening instrument including eight items specifically designed for the intensive care setting with two points: absent or present. The items include the assessment of: (1) consciousness (comatose, soporose, awake, or hypervigilant); (2) orientation; (3) hallucinations or delusions; (4) psychomotor activity; (5) inappropriate speech or mood; (6) attentiveness; (7) sleep-wake cycle disturbances; and (8) fluctuation of symptomatology. The maximum score is eight; scores of ≥4 indicate the presence of Delirium.
Death during hospital stay | single time point assessment during hospital stay (up to 4 weeks)
  assessment of number of patients with in-hospital death
Return to premorbid functional baseline | single time point assessment during hospital stay (up to 4 weeks)
  assessment of number of patients with return to premorbid functional baseline

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, PD Dr. med, Principal Investigator — Clinic for Intensive Care Medicine, University Hospital Basel
Locations (1):
- Clinic for Intensive Care Medicine, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Dittrich T, Marsch S, Egli A, Ruegg S, De Marchis GM, Tschudin-Sutter S, Sutter R. Predictors of infectious meningitis or encephalitis: the yield of cerebrospinal fluid in a cross-sectional study. BMC Infect Dis. 2020 Apr 23;20(1):304. doi: 10.1186/s12879-020-05022-6. PMID 32326881